CLINICAL TRIAL: NCT06865482
Title: Characteristics And Clinical Course Of Disease In Participants With Cardiomyopathy Associated With Friedreich Ataxia (CLARITY-FA)
Brief Title: Clinical Course Of Disease In Participants With FA-CM
Status: Recruiting | Type: Observational
Sponsor: Lexeo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: LX2006-02
Record Dates: First submitted 2025-02-18; First posted 2025-03-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Friedreich Ataxia; Cardiomyopathy
Keywords: Friedreich Ataxia; FA-CM; Cardiomyopathy; FA; Cardiac Disease
MeSH Terms: conditions — Friedreich Ataxia; Cardiomyopathies; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants ≥16 years of age with FA-CM: Participants ≥16 years of age with FA-CM
- Cohort 2: Participants ≥6 to <16 years of age with FA-CM: Participants ≥6 to <16 years of age with FA-CM

SUMMARY:
Characteristics and clinical course of disease In participants with cardiomyopathy associated with Friedreich Ataxia (CLARITY-FA)

DETAILED DESCRIPTION:
Study LX2006-02 is a prospective, longitudinal, low-intervention, multicenter, global study aimed at characterizing the nature and rate of cardiac disease progression in participants with genetically confirmed FA-CM. After completing at least 26 weeks in Study LX2006-02, participants who meet the eligibility criteria may have the opportunity to participate in an LX2006 interventional study and receive gene therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages ≥6 years at the time of signing the informed consent (and assent, if applicable).
* Diagnosis of FA, based on clinical phenotype and genotype (GAA expansion on both alleles or compound heterozygous), with onset of FA occurring at ≤25 years of age
* Confirmed left ventricular hypertrophy (LVH)
* Left ventricular ejection fraction ≥40%

Exclusion Criteria:

* Presence of other form(s) of CM contributing to heart failure (HF), clinically significant cardiac anatomic abnormality or congenital cardiac malformation, clinically significant coronary artery, uncorrected, hemodynamically significant primary structural valvular disease not due to CM
* Currently receiving intermittent or continuous intravenous (IV) inotrope infusion, presence of a ventricular assist device, or history of prior heart transplantation
* Contraindication to cMRI, participants <12 years of age who cannot complete the cMRI without sedation will instead undergo ECHOs and are exempt from this criterion.
* Prior organ transplantation
* Initiation of cardiac resynchronization therapy (CRT) within 6 months prior to screening.
* History of prior gene transfer or cell therapy.
* Poorly controlled diabetes (hemoglobin A1c ≥8%)
* Active hematologic or solid organ malignancy

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 65 participants with genetically confirmed FA-CM will be enrolled in the study with allocation by age categories and cohorts
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Characterize cardiac disease presentation and progression among participants | 26 weeks
  Change from baseline in left ventricular mass index (LVMi)

SECONDARY OUTCOMES:
Describe progression of left ventricular wall thickness (LVWT) among this population | 52 weeks
  Change from baseline
Describe progression of relative wall thickness (RWT) among this population | 52 weeks
  Change from baseline
Describe progression of relative wall mass (RWM) among this population | 52 weeks
  Change from baseline
Describe progression of left ventricular ejection fraction (LVEF) among this population | 52 weeks
  Change from baseline
Describe progression of left ventricular mass index (LVMi) among this population | 52 weeks
  Change from baseline
Describe progression of high sensitivity troponin I among this population | 52 weeks
  Change from baseline
Describe participant perception and clinician assessment of illness in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) | 52 weeks
  Change from baseline
Describe clinician assessment of illness in modified Friedreich Ataxia Rating Scale (mFARS) | 52 weeks
  Change from baseline
Describe participant perception of illness in Patient Global Impression of Severity (PGI-S) | 52 weeks
  Change from baseline
Describe participant perception of illness in Patient Global Impression of Change (PGI-C) | 52 weeks
  Change from baseline
Describe patterns of concomitant medication use among this population | 12 months
  Change from baseline in concomitant medication use, assessed using medication logs, electronic health records and patient self-report.
Describe changes to medication use among this population | 12 months
  Change from baseline in medication use, evaluated using prescription records, patient-reported medication, or clinician-reported changes.
Evaluate all-cause mortality | 12 months
  Time from baseline to the first occurrence of any event of death due to any cause
Evaluate major adverse cardiovascular events (MACE) | 12 months
  Time from baseline to the first occurrence of any MACE, defined as cardiovascular hospitalization/ambulatory visit, non-fatal stroke, non-fatal life-threatening arrhythmia, heart transplant, implantation of left ventricular assisted device (LVAD)
Cumulative measure of CV and non-CV related health care utilization (HRU) | 12 months
  Health care utilization will be assessed through a combination of:
  * Data captured via Electronic Data Capture (EDC) system (e.g., hospitalizations, emergency room visits, procedures),
  * Patient-reported information collected by the physician during scheduled study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Lexeo Clinical Trials, Study Director — Lexeo Therapeutics
Locations (10):
- United States (6):
  - University of California San Diego, La Jolla, California
  - University of South Florida, Tampa, Florida
  - Indiana University - Riley Children's Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
- Centre Hospitalier de Universite de Montreal (CHUM), Montreal, Quebec, Canada
- Motol University Hospital and the Second Faculty of Medicine, Prague, Czechia
- Institut de Cardiologie Hopital Pitie Salpetriere, Paris, France
- Hospital Univeritario Puerta de Hierro de Majadahonda, Majadahonda, Madrid, Spain